CLINICAL TRIAL: NCT01088880
Title: An Open-label, Exploratory Study to Establish the Safety and Efficacy of 3 Months Treatment With Canakinumab in Patients With Colchicine Resistant Familial Mediterranean Fever
Brief Title: Efficacy and Safety of Canakinumab in Patients With Colchicine Resistant Familial Mediterranean Fever
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CACZ885DTR01
Record Dates: First submitted 2010-03-16; First posted 2010-03-17 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: Familial Mediterranean Fever
Keywords: Familial Mediterranean Fever; canakinumab; colchicine resistance
MeSH Terms: conditions — Familial Mediterranean Fever | interventions — canakinumab

ARMS (1):
- Canakinumab (Experimental)
  Interventions: Drug: Canakinumab

INTERVENTIONS:
Drug: Canakinumab

SUMMARY:
Establish the safety and efficacy of 3 months treatment with canakinumab in patients with colchicine resistant Familial Mediterranean Fever.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between 12 and 75 years of age with active type 1 FMF disease (according to Tel-Hashomer criteria for diagnosis of FMF) despite colchicine therapy (1.5 to 2.0 mg/day).
* Patients who are intolerant to effective doses of colchicine (1.5 to 2 mg/day)
* Patients with demonstrated minimum 1 typical acute attack per month and genetic confirmation of diagnosis (with at least one of the known MEFV gene exon 10 mutations). Patients with manifested amyloidosis are excluded.
* Patients must have a historical data showing a frequency of at least 1 attack/month within the last 3 months before they can be enter the run-in period.
* Patients must have type 1 disease characterized by recurrent and short episodes of inflammation and serositis with an average of at least 1 documented acute FMF attack per month during the previous 6 months and lasting approximately 12 to 72 hours.
* Patients treated with IL-1 therapies must complete washout and have experienced at least 2 attacks since (e.g. Anakinra: 3 day washout; Rilonacept: 3 week washout)
* Patients treated with anti-TNF drugs must undergo appropriate washout. Prior to randomization, use of Etanercept must be discontinued for 4 weeks or use of Adalimumab or Infliximab must be discontinued for 8 weeks.
* Female subjects of childbearing potential must be using two acceptable methods of contraception
* Patients treated with Interferon therapies must complete 1 month washout period.

Exclusion Criteria:

* Patients with end-organ dysfunction due to amyloidosis (e.g. existing biopsy proven amyloidosis or proteinuria > 0.5 gram per day)
* Patients taking steroids within 1 month prior to baseline
* Presence or history of any other inflammatory rheumatic disease
* Positive PPD test (according to local guidance) where a latent or active TB infection cannot be excluded via Quantiferon (T-Spot or radiographic imaging if needed).
* Patients who are pregnant or lactating
* Presence of any active or chronic infection or any major episode of infection requiring hospitalization or treatment with i.v. antibiotics within 30 days or oral antibiotics within 14 days prior to screening
* History or a malignancy within the last 5 years, except for successfully excised squamous or basal cell carcinoma of the skin

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
To measure the effect of canakinumab on the frequency of FMF attacks defined as percentage of patients with at least 50% reduction in the attack frequency during 3 month treatment period. | 12 weeks

SECONDARY OUTCOMES:
To assess the effect of canakinumab with regard to percentage of patients with no attacks in month 3. | 12 weeks
To find the optimal dose of canakinumab for FMF in this population | 12 weeks
To assess changes in the severity (acute phase response and VAS evaluation of attack severity by patient) and duration of acute attacks during the treatment period | 12 weeks
To assess PK/PD properties of canakinumab by measuring canakinumab and IL-1beta levels before dosing
To evaluate the safety and tolerability of canakinumab by monitoring adverse events and patient discontinuations due to AE

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Istanbul Medical Faculty, Dept of Rheumatology, Capa, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Gul A, Ozdogan H, Erer B, Ugurlu S, Kasapcopur O, Davis N, Sevgi S. Efficacy and safety of canakinumab in adolescents and adults with colchicine-resistant familial Mediterranean fever. Arthritis Res Ther. 2015 Sep 4;17(1):243. doi: 10.1186/s13075-015-0765-4. PMID 26337145